CLINICAL TRIAL: NCT01572714
Title: Examining the Effects of Physical Activity Promotion, Fatigue Management Education, and Social Support Using a Telehealth Intervention Approach Among Adults With Multiple Sclerosis
Brief Title: Examining the Effects of a Telehealth Self-management Intervention in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Matthew Plow, Project Scientist, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-14-19
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Self Care; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Support Program (Active Comparator): The social support program will consist of 6 weekly, 1.25-hours, teleconference calls with 4 biweekly, 15 minute, follow-up one-to-one phone calls. Topics will include information on MS, disease modifying medications, preventive screening, community organizations, nutrition, cognitive problems, and hiring an aide.
  Interventions: Behavioral: Social Support Program
- Physical Activity Program (Active Comparator): The physical activity education program will consist of 3 weekly, 1.25-hours, teleconference calls with 4 biweekly, 15 minute, follow-up one-to-one phone calls. Subjects in this program will learn MS-specific benefits of physical activity, how to use a pedometer to self-monitor their progress for increasing physical activity levels, and learn strategies for maintaining their progress in the program.
  Interventions: Behavioral: Physical Activity Program
- Physical Activity Plus Fatigue (Active Comparator): The physical activity plus fatigue management education program will consist of 6 weekly, 1.25-hours, teleconference calls with 4 biweekly, 15 minute, follow-up one-to-one phone calls. Subjects in this program will learn MS-specific benefits of physical activity, how to use a pedometer to self-monitor their progress for increasing physical activity levels, and learn strategies for maintaining their progress in the program. In addition, subjects in this course will learn strategies to reduce fatigue, such as taking rest breaks and re-arranging workspace.
  Interventions: Behavioral: Physical Activity Plus Fatigue Management Education Program

INTERVENTIONS:
Behavioral: Social Support Program — The social support program will consist of 6 weekly, 1.25-hours, teleconference calls with 4 biweekly, 15 minute, follow-up one-to-one phone calls. Topics will include information on MS, disease modifying medications, preventive screening, community organizations, nutrition, cognitive problems, and hiring an aide.
  Other Names: Social support
  Arms: Social Support Program
Behavioral: Physical Activity Program — The physical activity education program will consist of 3 weekly, 1.25-hours, teleconference calls with 4 biweekly, 15 minute, follow-up one-to-one phone calls. Subjects in this program will learn MS-specific benefits of physical activity, how to use a pedometer to self-monitor their progress for increasing physical activity levels, and learn strategies for maintaining their progress in the program.
  Other Names: Physical Activity-only
  Arms: Physical Activity Program
Behavioral: Physical Activity Plus Fatigue Management Education Program — The physical activity plus fatigue management education program will consist of 6 weekly, 1.25-hours, teleconference calls with 4 biweekly, 15 minute, follow-up one-to-one phone calls. Subjects in this program will learn MS-specific benefits of physical activity, how to use a pedometer to self-monitor their progress for increasing physical activity levels, and learn strategies for maintaining their progress in the program. In addition, subjects in this course will learn strategies to reduce fatigue, such as taking rest breaks and re-arranging workspace.
  Other Names: Physical Activity +
  Arms: Physical Activity Plus Fatigue

SUMMARY:
The objective of this study is to conduct a randomized controlled trial to examine the effectiveness of a telehealth intervention that supports individuals in managing fatigue and increasing physical activity (PA) behavior in individuals with multiple sclerosis (MS). The hypothesis is that a fatigue management plus physical activity intervention will significantly improve fatigue, quality of life, physical function, and community integration.

DETAILED DESCRIPTION:
The long-term objective of this study is to use a telehealth intervention approach to reduce the devastating effects of the reciprocal relationship between fatigue and inactivity on quality of life and participation in life roles in people with multiple sclerosis (MS). Chronic fatigue and inactivity are common problems in persons with MS, and the reciprocal relationship between fatigue and inactivity may have negative synergistic effects on quality of life and participation in life roles. The proposed study is novel in that it represents a multi-disciplinary effort to merge two promising lines of MS research: fatigue management and PA promotion. The proposed fatigue management plus PA intervention (FM+) will consist of incorporating a modified teleconference version of Packer et al.'s empirically-tested Fatigue Management program with innovative, yet simple approaches to promote lifestyle PA by encouraging goal-setting and self-monitoring with a pedometer. Ambulatory individuals with MS will be recruited and randomized into one of three telehealth interventions: social support intervention, PA-only intervention, and FM+.

ELIGIBILITY:
Inclusion Criteria:

* A physician-confirmed diagnosis of MS

Exclusion Criteria:

* Exercise more than 90 minutes per week
* Pregnant
* Metabolic or cardiopulmonary disease that puts patient at high risk for engaging in a home exercise program (patients with controlled diabetes and high blood pressure will still be considered eligible)
* Four or more falls in the past 6 months
* Be able to walk 25 feet with or without a cane or walker
* Severe cognitive deficits
* A condition besides MS that had lead to hospitalization in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2011-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in physical activity levels | Each patient will be given the assessments at 3 points during the study, at baseline, interim test (an average of 12 weeks from baseline) and at posttest (an average of 24 weeks from baseline).
  Physical activity behavior will be measured with the Godin Leisure-Time Exercise Questionnaire and accelerometers.

SECONDARY OUTCOMES:
Changes from baseline in fatigue levels | Each patient will be given the questionnaire at 3 points during the study, at baseline, interim test (an average of 12 weeks from baseline) and at posttest (an average of 24 weeks from baseline).
  Fatigue will be measured with the Fatigue Impact Scale.
Changes from baseline in quality of life | Each patient will be given the questionnaires at 3 points during the study, at baseline, interim test (an average of 12 weeks from baseline) and at posttest (an average of 24 weeks from baseline).
  The SF-12, Multiple Sclerosis Impact Scale, and Community Participation Indicator (CPI) will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Plow, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Plow M, Motl RW, Finlayson M, Bethoux F. Response heterogeneity in a randomized controlled trial of telerehabilitation interventions among adults with multiple sclerosis. J Telemed Telecare. 2022 Oct;28(9):642-652. doi: 10.1177/1357633X20964693. Epub 2020 Oct 25. PMID 33100184
- [Derived] Plow M, Motl RW, Finlayson M, Bethoux F. Intervention Mediators in a Randomized Controlled Trial to Increase Physical Activity and Fatigue Self-management Behaviors Among Adults With Multiple Sclerosis. Ann Behav Med. 2020 Feb 21;54(3):213-221. doi: 10.1093/abm/kaz033. PMID 31595300
- [Derived] Plow M, Finlayson M, Liu J, Motl RW, Bethoux F, Sattar A. Randomized Controlled Trial of a Telephone-Delivered Physical Activity and Fatigue Self-management Interventions in Adults With Multiple Sclerosis. Arch Phys Med Rehabil. 2019 Nov;100(11):2006-2014. doi: 10.1016/j.apmr.2019.04.022. Epub 2019 Jun 21. PMID 31229528
- [Derived] Plow M, Finlayson M, Motl RW, Bethoux F. Randomized controlled trial of a teleconference fatigue management plus physical activity intervention in adults with multiple sclerosis: rationale and research protocol. BMC Neurol. 2012 Oct 16;12:122. doi: 10.1186/1471-2377-12-122. PMID 23072517